CLINICAL TRIAL: NCT05599334
Title: A Retrospective Observational Study of Adult Patients With Early-stage HER2-positive Breast Cancer, Treated With Neratinib as Extended Adjuvant Therapy in the Context of the European Early Access Program (NEAR)
Brief Title: A Retrospective Observational Study of Patients With Early-stage HER2-positive Breast Cancer, Treated With Neratinib
Acronym: NEAR
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS12501
Record Dates: First submitted 2022-02-10; First posted 2022-10-31 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Adjuvant Therapy; HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; Adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to describe the demographic and clinical profiles of patients with early-stage HER2+ breast cancer treated with neratinib as an extended adjuvant therapy as part of the Early Access Program (EAP) in Europe.

DETAILED DESCRIPTION:
Eligible patients were selected among those who had received at least one dose of neratinib in the context of the early access program conducted in Europe between 01 August 2017 and 31 December 2020 (the patient identification period) and residing in one of the five target following countries: Belgium, Croatia, France, Italy and Spain, which were part of the EAP. Patients were followed up until the end of the study observation period/study entry date (05 July 2022). As this study was retrospective, the decision to prescribe neratinib was taken prior to and independent of the proposal to select a patient for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion if they fulfill all of the following criteria:

  * Age ≥ 18 years at neratinib treatment initiation
  * Having received at least one initial dose of neratinib as an extended adjuvant therapy for the treatment of early-stage HER2+ breast cancer, in the context of the EAP in Europe, and between August 01, 2017 and December 31, 2020
  * Patients (or next of kin/legal representative, if applicable) who provide written informed consent or non-opposition.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all patients with early-stage HER2+ breast cancer having received at least one dose of neratinib as an extended adjuvant therapy in the context of the EAP in Europe between August 01, 2017 and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Suissa, Study Director — Pierre Fabre Médicament
Locations (25):
- Belgium (3):
  - Clinique Saint-Luc Bouge, Bouge
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Multidisciplinary Breast Unit of the University Hospital Leuven and Sint-Andries Hospital, Leuven
- University Hospital Center Zagreb, Department of Oncology, Breast Unit, Zagreb, Croatia
- France (3):
  - CHU Brest - Hôpital Morvan, Brest
  - Centre Bourgogne, Lille
  - Hopital Prive La Louviere, Lille
- Italy (5):
  - Ospedale San Donato- ASL 8 Arezzo, Arezzo
  - Ospedale Santa Croce, Fano
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Istituto Nazionale Tumori Fondazione G. Pascale, Dipartimento di Senologia Via Mariano Semmola, Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
- Spain (13):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Teknon Barcelona, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Instituto Valenciano de Oncología IVO, Servicio de Oncología Médica C/ Beltran Baguena, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital LLuís Alcanyís de Xàtiva, Valencia

REFERENCES:
- [Derived] Krizic M, Silovski T, Hoste G, Dedic Plavetic N, Romano O, Gonzalez Farre X, Cano Jimenez A, Guerrero Zotano A, Suissa J, Beghdad F, Dialla O, Zivanov M, De Laurentiis M. A Retrospective Observational Study of Extended Adjuvant Neratinib for HER2-Positive Early-Stage Breast Cancer in a European Early Access Program. Oncol Ther. 2025 Dec;13(4):1205-1224. doi: 10.1007/s40487-025-00392-w. Epub 2025 Oct 29. PMID 41160302

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib Arm: Eligible patients were selected among those who had received at least one dose of neratinib in the context of the EAP in Belgium, Croatia, France, Italy and Spain between 01 August 2017 and 31 December 2020 (the patient identification period).
Period: Overall Study
Arm/Group | Neratinib Arm
Started | 111
Completed | 108
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: The baseline characteristics have been analysed in 108 patients corresponding to the number of patients analysed in the Full Analysis Set
Groups:
- Neratinib Arm: Eligible patients were selected among those who had received at least one dose of neratinib in the context of the EAP in Europe between 01 August 2017 and 31 December 2020 (the patient identification period) and residing in one of the five target following countries: Belgium, Croatia, France, Italy and Spain, which were part of the EAP.
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 111 in the number of enrolled patients and 108 is the number of analysed patients in the FAS
  years
    number analyzed (Participants) | 108
    (all) | 49.2 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 111 in the number of enrolled patients and 108 is the number of analysed patients
  Participants
    number analyzed (Participants) | 108
    Female | 107
    Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The details of participants by ethnicity was not collected
Region of Enrollment [Number; unit: participants] — The number of enrolled participants is 111 for which the region has been analysed. of note, the region has not been analysed in the 108 analysed participants from the FAS. Population: The total number of participants of participants is 111 corresponding to the enrolled number of participants on which the disposition by country was analysed, as this was not analysed in the 108 patients corresponding to the FAS. Therefore, the distribution by region has been done out of 111 patients, and not out of 108 patients.
  participants
    Croatia | 35
    Spain | 24
    Italy | 21
    Belgium | 16
    France | 15

OUTCOME MEASURES:

1. Primary Outcome: Description of Age
Description: Age will be assessed in years = neratinib initiation date - date of birth
Time Frame: At baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
years | 49.2 (8.83)

2. Primary Outcome: Description of Gender
Description: Gender will be described in percentage of Male and Female among patients
Time Frame: At baseline
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  Female | 107
  male | 1

3. Primary Outcome: Description of BMI
Description: BMI will be assessed in kg/m2
Time Frame: At baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Kg/m²
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Kg/m² | 26.7 (5.36)

4. Primary Outcome: Menopausal Status
Description: Menopausal status will be described in percentage of Premenopausal, Perimenopausal, Postmenopausal, Surgical/other reason for amenorrhea
Time Frame: At baseline
Population: FAS
Measure: Number; unit: participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
participants
  premenopausal | 40
  perimenopausal | 5
  postmenopausal | 34
  surgical/other reason for amenorrhea | 11
  unavailable | 17
  Not applicable (Male) | 1

5. Primary Outcome: Comorbidities
Description: Comorbidities will be described in number and percentage of patients with at least one relevant comorbidity. Comorbidities were including but were not limited to: renal disease, liver disease, gastro-intestinal disorders, cardiovascular conditions, skin and subcutaneous disorders, diabetes (type I or II)
Time Frame: At baseline
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants | 26

6. Primary Outcome: HER2 Overexpression/Amplification Testing
Description: HER2 overexpression/amplification testing will be assessed by Immunohistochemistry (IHC), Fluorescence in situ hybridization (FISH), Chromogenic in situ hybridization (CISH)
Time Frame: At initial diagnosis
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  IHC 3+ (positive) | 81
  IHC 2+ (equivocal) | 24
  IHC no | 1
  Unknown | 2

7. Primary Outcome: Hormone Receptor Status
Description: Hormone receptor status will be described in percentage of patients with Estrogen receptor (ER) positive, Progesterone receptor (PR) positive, ER and PR negative
Time Frame: At initial diagnosis
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  Estrogen receptor (ER) positive | 91
  ER negative | 17
  progesterone receptor (PR) positive | 74
  PR negative | 34

8. Primary Outcome: Primary Tumor Location
Description: Primary tumor location will be described in percentage of patients with Left Breast cancer, Right Breast cancer
Time Frame: At initial diagnosis
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  Left breast | 47
  Right breast | 62

9. Primary Outcome: Primary Tumor Histology
Description: Primary tumor histology will be described in percentage of patients with Infiltrating ductal carcinoma, Infiltrating lobular carcinoma, Invasive carcinoma, Tubular, Other
Time Frame: At initial diagnosis
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  Infiltrating ductal carcinoma | 56
  Infiltrating lobular carcinoma | 3
  Invasive carcinoma | 43
  Other | 6

10. Primary Outcome: Histological Grade
Description: Histological grade will be described in percentage of patients with G1 Well differentiated, G2 Moderately differentiated, G3 Poorly differentiated, G4 Undifferentiated
Time Frame: At initial diagnosis
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  G1 Well differentiated | 5
  G2 Moderately differentiated | 34
  G3 Poorly differentiated | 54
  Unavailable | 15

11. Primary Outcome: Pathologic Stage (AJCC Classification) of Breast Cancer
Description: Higher is the stage worse is the cancer.
  Stage is defined as:
  1A: tumor (T) up to 2 cm + not spread outside the breast; no lymph nodes (LN).1B: Small clusters of cancer cells (CC) (0.2-2 mm) are found in LN, or T in the breast is < 2 cm and small clusters of CC are found in LN. 2A: No T in the breast, but cancer is in 1-3 axillary LN or in LN near the breastbone or T is 2 cm or smaller + has spread to 1-3 axillary LN or LN near the breastbone, or T is > 2 cm and < 5 cm and not spread to LN.2B: T is > 2 cm and < 5 cm and has spread to 1-3 axillary LN or LN near the breastbone, or T is > 5 cm and not spread to the LN. 3A: no T in the breast or the T is any size; cancer is found in 4-9 axillary LN or LN near the breastbone, or T is larger than 5 cm and small clusters of CC found in LN. 3B: T has spread to chest wall or breast skin + may have spread to up to 9 axillary LN. 3C: Cancer has spread to ≥10 axillary LN, LN near the collarbone, or LN near breastbone
Time Frame: At initial diagnosis
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib Arm
Number analyzed (Participants) | 108
Participants
  I | 21
  IIA | 17
  IIB | 29
  IIIA | 25
  IIIB | 5
  IIIC | 6
  Missing | 5

ADVERSE EVENTS:
Time Frame: From the baseline to the study entry date
Arm/Group | Neratinib Arm
All-Cause Mortality (participants affected / at risk) | 1/108
Serious Adverse Events (participants affected / at risk) | 12/108
Other Adverse Events (participants affected / at risk) | 10/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neratinib Arm (N=108)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Infected seroma (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Hepatic enzymze increased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neratinib Arm (N=108)
abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Decreased apetite (Metabolism and nutrition disorders) | 2 (2)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Dizziness (Nervous system disorders) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Oedema peripheral (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT05599334/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT05599334/SAP_001.pdf